CLINICAL TRIAL: NCT00374179
Title: A Phase 1, Escalating Dose Study of CT-322, a VEGFR-2 Antagonist, as Monotherapy in Patients With Advanced Solid Tumors and Non-Hodgkin's Lymphoma
Brief Title: CT-322 in Treating Patients With Advanced Solid Tumors and Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adnexus, A Bristol-Myers Squibb R&D Company (Industry)
Responsible Party: Medical Director, Adnexus, A Bristol-Myers Squibb R&D Company, Adnexus, A Bristol-Myers Squibb R&D Company
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-322.001
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — CT-322

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CT-322 — IV solution, weekly or bi-weekly

SUMMARY:
RATIONALE: CT-322 may stop the growth of solid tumors or non-Hodgkin's lymphoma by stopping blood flow to the cancer.

PURPOSE: This phase I trial is studying the side effects of CT-322 in treating patients with advanced solid tumors or non-Hodgkin's lymphoma.

ELIGIBILITY:
DISEASE CHARACTERISTICS

* Histologically proven advanced solid malignancy or NHL for which no standard therapy exists or for which standard therapy had failed
* No known brain or leptomeningeal disease
* No prior bone marrow transplant or stem cell rescue
* No histologically confirmed squamous non-small cell lung cancer (NSCLC) with central chest tumor(s) still in place

PATIENT CHARACTERISTICS

Age:

* 18 and over

Performance status:

* ECOG performance status ≤ 2

Life expectancy:

* > 3 months

Hematopoietic:

* ANC ≥ 1500/mL
* Platelets ≥ 100,000/mL
* Hemoglobin ≥ 9.0 g/dL; and not requiring transfusion > 1 unit/month

Hepatic:

* AST and ALT ≤ 2.5 x ULN; if liver function abnormalities are due to the underlying malignancy, then AST and ALT may be ≤ 5 x the ULN
* Bilirubin ≤ 1.5 x ULN
* aPTT and PT < 1.5 x ULN

Renal:

* Creatinine ≤ 1.5 x ULN; patients with serum creatinine > 1 x ULN must also have creatinine clearance (based on a 24-hour urine collection) ≤ 60 mL/min
* No proteinuria > 1+ on dipstick analysis; in the case of > 1+ dipstick proteinuria, a 24-hour urine collection for protein must be < 500 mg/24 hours
* Urinary protein/creatinine ratio < 1
* No glomerulonephritis

Cardiovascular:

* No coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, unstable angina, symptomatic congestive heart failure, severe uncontrolled hypertension, hemorrhagic or thrombotic stroke or any other CNS bleeding within the preceding 12 months
* LVEF normal by echocardiogram or MUGA within the past 12 months if there was prior exposure to anthracyclines or radiotherapy encompassing the heart

Immunologic:

* Not known to have human immunodeficiency virus (HIV), active hepatitis virus C (HVC), or active hepatitis virus B (HVB)

Other:

* Negative pregnancy test within 7 days prior to enrollment
* Not pregnant or breast feeding
* Fertile patients must agree to use effective contraception or commit to abstinence during the study period, or be surgically sterile
* No serious nonhealing wound, ulcer, or bone fracture
* Have the ability to understand and sign an informed consent document
* Be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* At least 4 weeks since prior biological or immunotherapy and recovered

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy and recovered
* At least 6 weeks for mitomycin C and nitrosoureas prior to study entry and recovered

Radiotherapy:

* At least 4 weeks since prior radiotherapy to a visceral organ and recovered

Surgery:

* At least 4 weeks since prior major or laparoscopic surgery and recovered
* At least 1 week since prior minor surgery

Other:

* No other concurrent anticancer therapy
* Not concurrently enrolled in another therapeutic clinical trial involving ongoing therapy
* No concurrent full dose, therapeutic anti-coagulation with warfarin or related oral anti-coagulants or unfractionated or low molecular weight heparins; low dose warfarin for catheter prophylaxis or acetylsalicylic acid ≤ 325 mg/day is acceptable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-08; Primary Completion 2008-11 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of CT-322 | Throughout the study

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of CT-322 in these patients; | Throughout the study
to assess whether antibodies to this drug develop in these patients; and | Throughout the study
to make a preliminary assessment of the biological activity of CT-322 to alter tumor growth. | Throughout the study

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Indiana University Cancer Center, Indianapolis, Indiana
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - Institute for Drug Development, San Antonio, Texas

REFERENCES:
- [Derived] Tolcher AW, Sweeney CJ, Papadopoulos K, Patnaik A, Chiorean EG, Mita AC, Sankhala K, Furfine E, Gokemeijer J, Iacono L, Eaton C, Silver BA, Mita M. Phase I and pharmacokinetic study of CT-322 (BMS-844203), a targeted Adnectin inhibitor of VEGFR-2 based on a domain of human fibronectin. Clin Cancer Res. 2011 Jan 15;17(2):363-71. doi: 10.1158/1078-0432.CCR-10-1411. Epub 2011 Jan 11. PMID 21224368